CLINICAL TRIAL: NCT00101582
Title: Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Weekly Doses of Palifermin (rHuKGF) for the Reduction of Oral Mucositis in Subjects With Advanced Head and Neck Cancer Receiving Radiotherapy With Concurrent Chemotherapy (RT/CT)
Brief Title: Palifermin for the Reduction of Oral Mucositis in Patients With Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20020402; NCT00963456 (obsolete NCT alias)
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Mucositis; Solid Tumors; Stomatitis; Head and Neck Cancer; Squamous Cell Carcinoma
Keywords: SCCHN; Palifermin; Mucositis; Oral Cavity; Oropharynx; Nasopharynx; Hypopharynx; Larynx; Mouth Pain; Mouth Sores; Radiation Therapy; Radiotherapy; Radiochemotherapy; Concurrent Chemotherapy; Xerostomia; Stomatitis; Mucosa; KGF; rHuKGF; Keratinocyte Growth Factor; HNC; Head and Neck Cancer; Oral Mucositis
MeSH Terms: conditions — Mucositis; Stomatitis; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Laryngeal Diseases; Oral Ulcer; Xerostomia | interventions — Fibroblast Growth Factor 7; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palifermin (Experimental): Participants received a single intravenous dose of palifermin at 180 μg/kg three days before the start of radiotherapy, and then 7 once weekly palifermin doses at the same dose level during a 7-week radiotherapy/chemotherapy course.
  Interventions: Drug: palifermin; Drug: cisplatin chemotherapy; Radiation: Radiotherapy
- Placebo (Placebo Comparator): Participants received a single IV dose of placebo three days before the start of radiotherapy, and then 7 once weekly placebo doses during a 7-week radiotherapy/chemotherapy course.
  Interventions: Drug: Placebo; Drug: cisplatin chemotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: palifermin
  Other Names: Kepivance; Recombinant Human Keratinocyte Growth Factor (rHuKGF)
  Arms: Palifermin
Drug: cisplatin chemotherapy — Commercially available cisplatin was administered as an intravenous infusion at a dose of 100 mg/m^2 on Days 1, 22, and 43.
Radiation: Radiotherapy — Radiotherapy was delivered in 200 cGy daily fractions, 5 days a week.

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of palifermin to determine if weekly doses can be safely administered to reduce the incidence (occurrence of), duration (length of time) and severity (amount of pain) of oral mucositis (painful sores in the mouth). Mucositis is a common side effect for patients receiving chemotherapy (cancer-killing drug) and radiotherapy (cancer-killing x-rays) for the treatment of head and neck cancer (HNC).

DETAILED DESCRIPTION:
This study consisted of 2 phases. The acute oral mucositis (OM) evaluation phase includes the time from randomization to the time of severe OM (WHO Grade 3 or 4) resolution (up to Week 12 or up to Week 15 for participants whose severe OM is not resolved at Week 12). In the acute OM evaluation phase, participants were randomized to receive either a single IV dose of palifermin or placebo at 180 μg/kg, 3 days before the start of radiotherapy, plus 7 once-weekly palifermin or placebo doses at the same dose level during a 7-week radio/chemotherapy course. In the long-term follow up phase, participants are followed until death, withdrawal of consent, or loss to follow-up. The long-term follow up phase is still ongoing.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically documented squamous cell carcinoma involving either the oral cavity, oropharynx, nasopharynx, hypopharynx, or larynx
* Newly diagnosed, locally advanced stage head and neck cancer (unresectable/unresected disease); American Joint Committee on Cancer [AJCC] Stage III, IVA or IVB amenable to radiotherapy with concurrent chemotherapy as the definitive treatment modality
* At least 50 Gray of radiation treatment to areas of the oral cavity/oropharynx mucosa that can be visualized
* Concurrent chemotherapy regimen of Cisplatin 100mg/m^2 on days 1, 22, and 43
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) less than or equal to 2
* Adequate hematologic, renal and hepatic function
* Negative pregnancy test by serum or urine
* Signed informed consent

Key Exclusion Criteria:

- Presence or history of any other primary malignancy (other than curatively treated in situ cervical cancer, or basal cell carcinoma of the skin without evidence of disease for greater than 3 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2005-08; Primary Completion 2007-09 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 03 August 2005 (first participant enrolled) to 11 September 2007 (last participant's last visit at 4 months of follow-up) at 46 study centers in the United States, Canada, and Europe At the time of this report, the long-term safety follow-up period is ongoing.
Groups:
- Placebo: Participants received a single intravenous (IV) dose of placebo three days before the start of radiotherapy, and then 7 once weekly placebo doses during a 7-week radiotherapy/chemotherapy course. Chemotherapy consisted of 100 mg/m^2 cisplatin administered by IV infusion on Days 1, 22, and 43.
- Palifermin: Participants received a single intravenous dose of palifermin at 180 μg/kg three days before the start of radiotherapy, and then 7 once weekly palifermin doses at the same dose level during a 7-week radiotherapy/chemotherapy course. Chemotherapy consisted of 100 mg/m^2 cisplatin administered by IV infusion on Days 1, 22, and 43.
Period: Overall Study
Arm/Group | Placebo | Palifermin
Started | 94 | 94
Received Study Drug | 91 | 94
Completed | 83 (Participants who completed the acute oral mucositis evaluation phase) | 79 (Participants who completed the acute oral mucositis evaluation phase)
Not Completed | 11 | 15
Not completed — Ineligibility determined | 0 | 1
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Death | 3 | 5
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Palifermin | Total
Number analyzed (Participants) | 94 | 94 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (8.3) | 55.5 (8.6) | 55.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 80 | 79 | 159
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 90 | 83 | 173
  Black | 2 | 7 | 9
  Hispanic | 2 | 3 | 5
  American Indian/ Alaska Native | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: kilograms] — Data available for 91 and 94 participants in each treatment group respectively.
  kilograms | 71.8 (15.7) | 74.5 (16.4) | 73.2 (16.1)
Disease Stage [Number; unit: participants] — American Joint Committee on Cancer staging system.
  participants
    Stage III | 29 | 26 | 55
    Stage IV A | 54 | 60 | 114
    Stage IV B | 11 | 8 | 19
Tumor Site [Number; unit: participants]
  Oral Cavity | 9 | 5 | 14
  Oropharynx | 51 | 55 | 106
  Nasopharynx | 3 | 4 | 7
  Larynx | 9 | 16 | 25
  Hypopharynx | 22 | 14 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe (Grade 3 or 4) Oral Mucositis
Description: Participants underwent evaluations of oral mucosal (OM) surfaces (mucositis assessments) 2 times weekly throughout radio/chemotherapy, and 2 times weekly thereafter until severe OM returned to grade ≤ 2 or until Week 15. During each evaluation, the following anatomical areas were assessed: upper lip; lower lip; right cheek; left cheek; right ventral & lateral tongue; left ventral & lateral tongue; floor of the mouth; hard palate; soft palate. A trained evaluator documented the findings using the World Health Organization (WHO) oral toxicity scale according to the following: Grade 0 = None; Grade 1 = Soreness, erythema; Grade 2 = Erythema, ulcers, ability to eat solids; Grade 3 = Ulcers, requires liquid diet; Grade 4 = Alimentation not possible.
Time Frame: Up to Week 15
Population: The Full Analysis Set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 94 | 94
participants
  Yes | 62 | 51
  No | 29 | 43
  Unknown | 3 | 0
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Sample size calculations were based on the number of participants needed to detect, with 90% power and 5% type 1 error rate, at least a 25% difference in the incidence of severe OM between the treatment groups. A 25% absolute reduction in the incidence of severe OM from the placebo group was considered by investigators as clinically meaningful in this clinical setting; Test type: Superiority or Other; p = 0.0410, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association. Participants having no assessment were assumed as having WHO grade 3 or 4 oral mucositis in hypothesis testing; Stratified by disease stage (III versus IV) and primary anatomical tumor location (oral cavity / oropharynx vs. nasopharynx vs. hypopharynx / larynx); Chi-Square Statistic = 4.1764

2. Secondary Outcome: Duration of Severe (WHO Grade 3 or 4) Oral Mucositis
Description: The duration of severe oral mucositis (OM) was calculated as the number of days from the onset of severe OM (first time a WHO grade 3 or 4 was observed) to the day when severe OM was resolved (first time WHO grade 2 or less was observed after last WHO grade 3 or 4). Durations of 0 days were assigned to those participants who did not experience any WHO grade 3 or 4 during the study.
Time Frame: Up to 15 weeks
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 94 | 94
days | 26.0 [0.0 to 50.0] | 5.0 [0.0 to 40.0]
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.0160, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for mean score difference; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 5.8002
Statistical Analysis 2: Comparison: Placebo vs Palifermin; To protect the overall type 1 error, the Hochberg procedure was used to adjust for multiple statistical testing of the secondary efficacy endpoints; Test type: Superiority or Other; p = 0.1122, Cochran-Mantel-Haenszel — Adjusted p-value was based on Hochberg procedure to control for the Type 1 error

3. Secondary Outcome: Time to Onset of Severe (WHO Grade 3 or 4) Oral Mucositis
Description: Time to onset of severe (WHO Grade 3 or 4) oral mucositis (OM) was analyzed using the Kaplan-Meier procedure.
  Participants without an assessed event by the end of the acute OM evaluation phase were censored at the date of last assessment for severe OM.
Time Frame: Up to 15 weeks
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 94 | 94
days | 35.0 [22.0 to NA] — Could not be estimated due to the low number of events | 47.0 [27.0 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.0261, Stratified Log-Rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.6603, 95% CI 2-sided [0.4546 to 0.9592] — Hazard ratio of palifermin over placebo based on Stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.1566, Stratified Log-Rank test — Adjusted p-value was based on Hochberg procedure to control for the Type 1 error

4. Secondary Outcome: Number of Participants With Xerostomia at Month 4 (Grade 2 or Higher)
Description: The number of participants with grade 2 or higher xerostomia (dryness of the oral mucosa) at the Month 4 visit, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Dry Mouth/Xerostomia scale.
Time Frame: Month 4
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 94 | 94
participants
  Yes | 57 | 37
  No | 19 | 31
  Unknown | 18 | 26
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.0463, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association. Participants having no assessment were assumed to have the event; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 3.9715
Statistical Analysis 2: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.2314, Cochran-Mantel-Haenszel — Adjusted p-value was based on Hochberg procedure to control for the Type 1 error

5. Secondary Outcome: Patient-Reported Mouth and Throat Soreness Score
Description: The average patient-reported mouth and throat soreness (MTS) score as reported on question 3 of the Oral Mucositis Weekly Questionnaire for Head and Neck Cancer [OMWQ-HN]): "How much mouth and throat soreness did you experience in the past 24 hours?" Participants answered on a scale from 0 (no soreness) to 4 (extreme soreness).
  For each participant, an average patient-reported mouth and throat soreness score was calculated by dividing the sum of the MTS scores at each assessment by the total number of assessments.
Time Frame: Assessed twice a week for up to 15 weeks.
Population: The Patient Reported Outcome-evaluable analysis set included all randomized patients with a valid Baseline assessment for MTS question 3 of the OMWQ-HN and either:
  * At least 1 completed assessment each week for MTS up to withdrawal/Week 8, whichever came first, or
  * 70% or greater overall compliance for MTS until withdrawal/Week 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 88 | 89
units on a scale | 1.86 (0.65) | 1.66 (0.73)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.0712, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for mean score difference using modified ridit score; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 3.2548
Statistical Analysis 2: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.2849, Cochran-Mantel-Haenszel — Adjusted p-value was based on Hochberg procedure to control for the Type 1 error

6. Secondary Outcome: Total Dose of Opioid Analgesics Used for Mucositis Within 15 Weeks
Description: The total dose of opioid analgesics (mg of intravenous [IV] morphine equivalents) used by all participants.
  Participants with at least one reported administration of opioid analgesic (parenteral, peroral or transdermal) were considered to have received opioid analgesics. The total dose of opioid analgesics is the sum of all opioid analgesic administrations that have been converted to morphine equivalents.
Time Frame: Up to 15 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg of IV morphine equivalents
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 94 | 94
mg of IV morphine equivalents | 1219.55 (1769.29) | 1243.31 (2700.28)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.2384, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for mean score difference using modified ridit score; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 1.3901
Statistical Analysis 2: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.6835, Cochran-Mantel-Haenszel — Adjusted p-value was based on Hochberg procedure to control for the Type 1 error

7. Secondary Outcome: Number of Participants With Unplanned Breaks in Cisplatin Chemotherapy Treatment
Description: Cisplatin was administered on Days 1, 22, and 43. An unplanned break in cisplatin refers to a delay of ≥ 5 days from the scheduled Day 22 or Day 43 cisplatin administration or a discontinuation of cisplatin for any reason.
Time Frame: During the 7 weeks of chemotherapy treatment
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 94 | 94
participants | 42 | 49
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.3417, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 0.9039
Statistical Analysis 2: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.6835, Cochran-Mantel-Haenszel — Adjusted p-value was based on Hochberg procedure to control for the Type 1 error

8. Secondary Outcome: Number of Participants With Unplanned Breaks in Radiotherapy
Description: Participants with a duration of 5 days or more without an administration of radiotherapy or who discontinue radiotherapy prior to completion of planned radiotherapy were considered to have an unplanned break in radiotherapy.
Time Frame: During the 7 weeks of radiotherapy
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 94 | 94
participants | 11 | 13
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.9587, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 0.0027
Statistical Analysis 2: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.9587, Cochran-Mantel-Haenszel — Adjusted p-value was based on Hochberg procedure to control for the Type 1 error

ADVERSE EVENTS:
Time Frame: Approximately 8 weeks
Description: The table of Other Adverse Events summarizes non-serious occurrences of adverse events that exceeded a 5% frequency in either treatment arm.
Groups:
- Placebo: Participants received a single intravenous (IV) dose of placebo three days before the start of radiotherapy, and then 7 once weekly placebo doses during a 7-week radiotherapy/chemotherapy course.
Arm/Group | Placebo | Palifermin
Serious Adverse Events (participants affected / at risk) | 25/91 | 35/94
Other Adverse Events (participants affected / at risk) | 81/91 | 89/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | Palifermin (N=94)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 1 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 1 | 4
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchitis acute (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 2
Clostridial infection (Infections and infestations) | 0 | 1
Colitis pseudomembranous (Infections and infestations) | 1 | 1
Infected epidermal cyst (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pulmonary sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Device occlusion (Injury, poisoning and procedural complications) | 0 | 1
Injury asphyxiation (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin abnormal (Investigations) | 0 | 1
Blood creatinine abnormal (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
Blood lactate dehydrogenase abnormal (Investigations) | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood sodium abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 5
White blood cell count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 9 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peritoneal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Syncope vasovagal (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 1
Cryptogenic organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | Palifermin (N=94)
Anaemia (Blood and lymphatic system disorders) | 32 | 21
Leukopenia (Blood and lymphatic system disorders) | 11 | 21
Neutropenia (Blood and lymphatic system disorders) | 6 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2
Tinnitus (Ear and labyrinth disorders) | 7 | 11
Constipation (Gastrointestinal disorders) | 24 | 31
Diarrhoea (Gastrointestinal disorders) | 14 | 7
Dry mouth (Gastrointestinal disorders) | 5 | 9
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Dysphagia (Gastrointestinal disorders) | 19 | 27
Nausea (Gastrointestinal disorders) | 42 | 46
Odynophagia (Gastrointestinal disorders) | 5 | 9
Oesophagitis (Gastrointestinal disorders) | 0 | 5
Oral pain (Gastrointestinal disorders) | 3 | 9
Vomiting (Gastrointestinal disorders) | 24 | 24
Asthenia (General disorders) | 5 | 4
Fatigue (General disorders) | 20 | 21
Malaise (General disorders) | 1 | 5
Oedema peripheral (General disorders) | 4 | 6
Pyrexia (General disorders) | 19 | 16
Candidiasis (Infections and infestations) | 14 | 11
Oral candidiasis (Infections and infestations) | 11 | 17
Oral fungal infection (Infections and infestations) | 6 | 5
Radiation skin injury (Injury, poisoning and procedural complications) | 13 | 25
Blood creatinine increased (Investigations) | 4 | 7
Weight decreased (Investigations) | 26 | 25
Anorexia (Metabolism and nutrition disorders) | 10 | 12
Dehydration (Metabolism and nutrition disorders) | 12 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 19
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5
Dizziness (Nervous system disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 7 | 18
Headache (Nervous system disorders) | 5 | 10
Anxiety (Psychiatric disorders) | 8 | 9
Depression (Psychiatric disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 10 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 6
Dermatitis (Skin and subcutaneous tissue disorders) | 10 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 5
Flushing (Vascular disorders) | 0 | 6
Hypertension (Vascular disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits sponsor a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Sponsor may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, investigator agrees not to publish any results before the first multi-center publication.